CLINICAL TRIAL: NCT04941625
Title: Risk of Acute Kidney Injury in Patients Undergoing Cytoreductive Surgery and Hyperthermic Intra-peritoneal Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chao-Yu Chen, Associated Professor, Chang Gung Memorial Hospital
Other Study IDs: 201701400A3
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Acute Kidney Injury
Keywords: Peritoneal malignancy; hyperthermic intraperitoneal chemotherapy; acute kidney injury; renal insufficiency
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples were evaluated using standard laboratory methods. The serum-cystatin C concentration and urine-NGAL in non-AKI and AKI groups are measured pre-operative day, post-operative 2h, 24h, 48h, 72h and day 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-AKI: patients do not have post-HIPEC AKI
  Interventions: Diagnostic Test: serum cystatin C; Diagnostic Test: serum beta-microglubulin; Diagnostic Test: urine
- AKI: patients have post-HIPEC AKI
  Interventions: Diagnostic Test: serum cystatin C; Diagnostic Test: serum beta-microglubulin; Diagnostic Test: urine

INTERVENTIONS:
Diagnostic Test: serum cystatin C — blood sampling
Diagnostic Test: serum beta-microglubulin — blood sampling
Diagnostic Test: urine — neutrophil gelatinase-associated lipocalin

SUMMARY:
Background: Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) is an emerging surgical procedure for peritoneal carcinomatosis. Despite the survival benefits from HIPEC, complications have been reported with major morbidity and mortality. Acute kidney injury (AKI) is one of the major complications. To date, there is no adequate biomarker to predict the risk of AKI after HIPEC and monitor the renal prognosis after HIPEC-related AKI.

Aims:

1. Establish a HIPEC cohort database, including retrospective data and prospective database
2. Identify the incidence of AKI after HIPEC and the severity
3. Identify the biomarker to predictive HIPEC-related AKI and monitor renal prognosis. Understand the risk factors for AKI post- HIPEC helps improve pre-operative patient selection and optimization, facilitate tailoring of chemotherapy, and foster closer peri-operative monitoring and fluid management in at-risk patients.

Methods:

1. Patients with the peritoneal carcinomatosis, planning to receive HIPEC and agree to participate the study will be recruited.
2. Retrospective analyze the renal prognosis of patients with HIPEC procedure and identify the clinical and biochemistry risk factors of HIPEC-related AKI
3. Prospective collect the information of patients who are enrolled into this study. The information includes clinical information, biochemistry, electrolyte, and novel biomarkers of body fluids (blood, and urine). The samples of body fluids will be collected on pre-operative day, post-operative 2h, 24h, 48h, 72h and day 7. Patients with or without post-HIPEC AKI will be analyzed.

Hypothesis:

1. Peri-operative dehydration and cisplatin-based regimen are the major risk factors to cause AKI.
2. The novel biomarker, high peri-operative urine NGAL and serum cystatin C, β2 Microglobulin are the predictive markers of HIPEC- related AKI.

DETAILED DESCRIPTION:
Introduction Peritoneal carcinomatosis (PC) is a serious oncological condition in patients with metastatic malignancy, for which cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CRS/HIPEC) has become the treatment of choice. In this procedure, chemotherapeutic drugs are introduced intraoperatively into the peritoneal cavity at temperature 41-43 °C. The abdominal cavity is perfused for about 60-90 minutes, thereby exposing potential microscopic residual cancer cells directly to the synergistic effects of hyperthermia (Sugarbaker 2016). In highly selected patients with colorectal cancer, CRS/HIPEC has shown benefits in disease-free and overall survival compared to systemic chemotherapy alone, with a 5-year survival rate of up to 45% for patients with no residual tumor after completing CRS. Furthermore, in patients with PMP receiving CRS/HIPEC, the survival rate beyond 10 years has been reported to reach 63% (Yan, Stuart et al. 2006, Verwaal, Bruin et al. 2008).

CRS/HIPEC is an aggressive treatment modality, often associated with high-grade complications. Recent publications have reported morbidity and mortality rates of 2.5-25% and 1.5-11%, respectively, with renal toxicity and bone marrow failure accounting for most causes of systemic toxicity (Ihemelandu, McQuellon et al. 2013, Wang, Chen et al. 2017). Acute kidney injury (AKI) is a serious morbidity that is associated with a greater duration of hospitalization, higher risk of mortality and increased risk of progressive chronic kidney disease. It has been described after the administration of HIPEC with cisplatin, with the quoted incidence of major renal toxicity ranging from 1.3-5.9% (Sin, Chia et al. 2017).

Renal toxicity of HIPEC Chemotherapy effect Cisplatin, a platinum-based anticancer agent, exerts its cytotoxic effect by binding and cross-linking DNA. It has been utilized as a cornerstone in many HIPEC protocols at variable doses for the treatment of tumors with PC, including primary peritoneal neoplasms, sarcomas, and gynecological tumors. Cisplatin-induced nephrotoxicity is a complex process involving acute cytotoxicity to tubular epithelium, followed by inflammatory cell infiltration and fibroproliferative changes. A recent pharmacokinetic study of this regimen yielded a cisplatin perfusate-to-blood area under the curve ratio of 6.28. These data indicate the absorption of cisplatin into the circulation during HIPEC, hence systemic complications cannot be excluded. Western literatures reported that 4-6% incidence of renal toxicity among patients who underwent HIPEC using cisplatin at variable doses and combinations (Hakeam, Breakiet et al. 2014). However, higher incidence of renal toxicity was reported by Singapore. Tan et al reported that among the 47 patients, 19 (40.4%) experienced post-operative AKI, of which 5 (8.5%) developed grade 3 and 4 impairment. Two (4.3%) required long-term dialysis.

In addition, mitomycin and doxorubicin which are also often used as HIPEC regimens, are also known nephrotoxins (Hakeam, Breakiet et al. 2014).

Comorbidity effect Preexisting kidney damage, hypomagnesemia and concomitant use of other nephrotoxic agents may potentiate the development of renal impairment. Other factors associated with nephrotoxicity were possible lower intraoperative urine output, and diabetes mellius (Yan, Stuart et al. 2006, Hakeam, Breakiet et al. 2014).

Biomarker of renal toxicity The traditional diagnosis of AKI involves measurements of surrogate markers of the reduced glomerular filtration rate (GFR), such as a rise in serum creatinine levels and/or a reduction in urine output. However, measurement of serum creatinine levels has limitation as a screening test in the early stages of AKI (Schiffl and Lang 2012). The emergence of numerous renal tubular damage-specific biomarkers offers an opportunity to diagnose AKI at an early time point, to facilitate differential diagnosis of structural and functional AKI, and to predict the outcome of established AKI. The reported potential biomarkers are cystatin C and NGAL (neutrophil gelatinase-associated lipocalin).

Cystatin C Serum cystatin C concentration has been described in numerous studies as being superior to serum creatinine for assessment of glomerular filtration rate. Adding serum cystatin C to the combi¬nation of serum creatinine and albuminuria improved the predictive accuracy of a model of all-cause mortal¬ity and ESRD. Elevated serum levels of cystatin C are also associated with renal and cardiovascular complica¬tions.

NGAL Serum and urinary levels of neutrophil gelatinase-associated lipocalin (NGAL) are elevated in several renal pathologies, including chronic glomerular disease, autosomal dominant polycystic kidney disease, and AKI. Elevated plasma NGAL was also suggested to be an excellent biomarker of com-plications associated with kidney disease, such as cardiovascular disease, and to be associated with progression as well as inhibition of tumor growth.

Beta-2 microglobulin β2 Microglobulin is a non-glycosylated protein. In the system, it possesses the negative charge. β2 Microglobulin is a component of MHC class 1 molecules, which are present on almost all cells of the body except red blood cells. β2 Microglobulin is generally required for the transport of MHC class I heavy chains from the endoplasmic reticulum to the cell surface. β2 Microglobulin is filtered by the glomerulus, absorbed and catabolised by the proximal tubules. Clinically the appearance of significant amount of this protein in urine is one of the earliest sign of almost all renal diseases. Serum creatinine is affected by factors other than GFR, in particular muscle mass and meat intake. β2 Microglobulin is released at constant rate in normal subjects, readily filters through the glomerular capillary wall, over 99.9% being reabsorbed and catabolised in proximal tubules with virtually no return of the filtered protein to the circulation. β2 Microglobulin is therefore theoretically a highly suitable biomarker of renal dysfunction.

Preliminary findings of HIPEC in Chang-Gung Memorial Hospital at Chiayi In the report of our preliminary data, the grade 3 complications were 30.7% in the very early cases and 12.4% after establishing multi-disciplinary teamwork (MDT) (Wang, Chen et al. 2017). We noted a trend of AKI in patients who underwent HIPEC with cisplatin. Permanent kidney injury was noted in two patients and transient AKI was noted in three cases in this database (2015/4-2016/12). Further two patients suffered from grade 3-4 AKI was also noted in 2017 even under MDT care.

Aims Previous studies mostly discuss the clinical risk factors of renal toxicity. Literature of biomarker related to HIPEC-related AKI is sparse. Herein, firstly, we aim to establish a HIPEC cohort database and retrospectively study the patients suffered from HIPEC-related AKI and identify the clinical risk factors and the renal prognosis. Furthermore, we will recruit blood, and urine samples to identify the novel biomarker to predictive HIPEC-related AKI and monitor renal prognosis. This can help to identify the risk factors for AKI and improve pre-operative patient's selection, facilitate tailoring of chemotherapy, and foster closer peri-operative monitoring and fluid management in high-risk patients.

Hypothesis

1. After retrospective chart review, peri-operative dehydration during operation (massive bleeding, prolong surgery with hyperthermia, etc) after HIPEC and cisplatin-based regimens are the major risk factor to cause AKI.
2. The novel biomarker, higher pre-operative urine NGAL and serum cystatin C, β2 Microglobulin are the predictive markers of patients who will have the peri-operative dehydration and correlate with HIPEC -related AKI.

Aim 1. To establish a HIPEC cohort database and retrospectively study the patients suffered from HIPEC-related AKI and identify the clinical risk factors and the renal prognosis.

Aim 2. To identify the novel biomarker (urine NGAL and serum cystatin C) to predictive HIPEC-related AKI and monitor renal prognosis.

Study design:

Aim 1. A single institution (Chang Gung Memorial Hospital at Chiayi), retrospective study Aim 2. Prospective cohort study to validate Aim 1. Clinical data, blood and urine samples should be collected.

Number of patients:

Aim 1. Chart review of patients who receiving HIPEC procedure from 2015/4-2018/12. The estimated case numbers are 180 cases. (100 cases of 2015/4-2017/9 plus estimated 80 cases from 2017/10-2017/12) Aim 2. Prospective collection of clinical data of 150 patients (estimated 50-60 cases /year).

Collect data:

Patient age, gender, cancer type, disease status (primary or recurrent), grade of differentiation, histology type, tumor burden (peritoneal carcinomatosis index), date of diagnosis/recurrence, site/pattern of recurrence, performance states, date of operation date, HIPEC parameters (chemotherapy regimens, perfusate, cytoreduction time, duration, and temperatures), peri-operative fluid status, pre-operative imaging date and types (CT or MRI, with or without contrast which is related to renal function), and date of death or lost to follow-up.

Routinely blood data are collected (CBC/DC, serum creatinine, BUN, liver function test, albumin, electrolyte, sugar, osmolarity…) on pre-operative, post-HIPEC 2hr, post-HIPEC 24 hours, 48 hours, 72 hours, day 7, and day 30.

Samples collection:

Blood and urine samples were evaluated using standard laboratory methods. The serum-cystatin C concentration and urine-NGAL in non-AKI and AKI groups are measured pre-operative day, post-operative 2h, 24h, 48h, 72h and day 7.

Statistic analysis:

The data will be analyzed by the SPSS 17·0 statistical package. Chi-square test and t-test for single variate analysis will be used to evaluate the association between covariates. Survival curves (cancer-specific survival [CSS] and recurrence-free survival [RFS]) will be generated using the Kaplan-Meier method. Multivariate analysis by cox stepwise forward regression will be used. Generalized estimating equation (GEE) will be used for those repeated measured data. Their hazard ratios (HR) and 95% confidence intervals (CI) will be calculated. All tests will be two-sided, and p values of < 0·05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receive HIPEC treatment
2. Age >20 y/o, < 75 y/o

Exclusion Criteria:

1. baseline creatinine >1.5 or GFR < 50
2. AST, ALT, bilirubin > 3x normal upper limit
3. one kidney or previous renal surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receive HIPEC treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 1 week
  RIFLE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yu Chen, MD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Chang Gung Memorial Hospital, Chiayi, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data entry personnel will enter de-identified data of the patients as per the datasheet

REFERENCES:
- [Background] Hakeam HA, Breakiet M, Azzam A, Nadeem A, Amin T. The incidence of cisplatin nephrotoxicity post hyperthermic intraperitoneal chemotherapy (HIPEC) and cytoreductive surgery. Ren Fail. 2014 Nov;36(10):1486-91. doi: 10.3109/0886022X.2014.949758. Epub 2014 Aug 26. PMID 25155314
- [Background] Ihemelandu CU, McQuellon R, Shen P, Stewart JH, Votanopoulos K, Levine EA. Predicting postoperative morbidity following cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (CS+HIPEC) with preoperative FACT-C (Functional Assessment of Cancer Therapy) and patient-rated performance status. Ann Surg Oncol. 2013 Oct;20(11):3519-26. doi: 10.1245/s10434-013-3049-8. Epub 2013 Jun 8. PMID 23748607
- [Background] Schiffl H, Lang SM. Update on biomarkers of acute kidney injury: moving closer to clinical impact? Mol Diagn Ther. 2012 Aug 1;16(4):199-207. doi: 10.1007/BF03262209. PMID 22650449
- [Background] Sin EI, Chia CS, Tan GHC, Soo KC, Teo MC. Acute kidney injury in ovarian cancer patients undergoing cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy. Int J Hyperthermia. 2017 Sep;33(6):690-695. doi: 10.1080/02656736.2017.1293304. Epub 2017 Mar 5. PMID 28540777
- [Background] Sugarbaker PH. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in the management of gastrointestinal cancers with peritoneal metastases: Progress toward a new standard of care. Cancer Treat Rev. 2016 Jul;48:42-9. doi: 10.1016/j.ctrv.2016.06.007. Epub 2016 Jun 16. PMID 27347669
- [Background] Verwaal VJ, Bruin S, Boot H, van Slooten G, van Tinteren H. 8-year follow-up of randomized trial: cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy in patients with peritoneal carcinomatosis of colorectal cancer. Ann Surg Oncol. 2008 Sep;15(9):2426-32. doi: 10.1245/s10434-008-9966-2. Epub 2008 Jun 3. PMID 18521686
- [Background] Wang TY, Chen CY, Lu CH, Chen MC, Lee LW, Huang TH, Hsieh MC, Chen CJ, Yu CM, Chuang HC, Liao TT, Tseng CW, Huang WS. Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy for peritoneal malignancy: preliminary results of a multi-disciplinary teamwork model in Asia. Int J Hyperthermia. 2018 May;34(3):328-335. doi: 10.1080/02656736.2017.1337238. Epub 2017 Jun 23. PMID 28562119
- [Background] Yan TD, Stuart OA, Yoo D, Sugarbaker PH. Perioperative intraperitoneal chemotherapy for peritoneal surface malignancy. J Transl Med. 2006 Apr 10;4:17. doi: 10.1186/1479-5876-4-17. PMID 16606461